CLINICAL TRIAL: NCT02553889
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Study of the Safety, PK, and PD of Multiple Doses of ISIS 416858 (ISIS-FXI RX), Administered Subcutaneously to Patients With End-Stage Renal Disease on Hemodialysis
Brief Title: A Study of Safety, PK, & PD of ISIS 416858 Administered Subcutaneously to Patients With End-Stage Renal Disease on Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ISIS 416858 CS4
Record Dates: First submitted 2015-09-14; First posted 2015-09-18 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: End-stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ISIS 416858

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PK Cohort (Experimental): A 4-week screening period followed by a 4-week treatment period followed by a 6-week post-treatment evaluation period. Treatment period includes 1 dose of 300 mg ISIS 416858 on Day 1 and again on Day 29. Both doses of Study Drug will be administered subcutaneously (SC).
  Interventions: Drug: ISIS 416858
- Cohort A (Placebo Comparator): Patients in Cohort A will be randomized to receive either 200 mg ISIS 416858 or placebo. A 2:1 ratio will be used.
  For Cohort A, the study will include a 4-week screening period and a 12-week treatment period followed by a 12-week post-treatment evaluation period.
  Cohort A will receive Study Drug (ISIS 416858 or placebo) twice a week during the first 2 weeks, followed by once weekly for the remaining 10 weeks of the treatment period. All doses of Study Drug will be administered subcutaneously (SC) 10 minutes after completion of the hemodialysis treatment.
  Interventions: Drug: ISIS 416858; Drug: Placebo
- Cohort B (Placebo Comparator): Patients in Cohort B will be randomized to receive either 300 mg ISIS 416858 or placebo. A 2:1 ratio will be used.
  For Cohort B, the study will include a 4-week screening period and a 12-week treatment period followed by a 12-week post-treatment evaluation period.
  Cohort B will receive Study Drug (ISIS 416858 or placebo) twice a week during the first 2 weeks, followed by once weekly for the remaining 10 weeks of the treatment period. All doses of Study Drug will be administered subcutaneously (SC) 10 minutes after completion of the hemodialysis treatment.
  Interventions: Drug: ISIS 416858; Drug: Placebo

INTERVENTIONS:
Drug: ISIS 416858 — subcutaneous injection
  Other Names: ISIS-FXI Rx; BAY2306001; IONIS-FXI Rx
Drug: Placebo — subcutaneous injection
  Other Names: 0.9% sterile saline
  Arms: Cohort A; Cohort B

SUMMARY:
Evaluation of safety, tolerability, PK and PD of ISIS 416858 in patients with end-stage renal disease (ESRD) receiving chronic hemodialysis.

DETAILED DESCRIPTION:
Evaluation of Safety, PK and PD of ISIS 416858 in patients with end-stage renal disease (ESRD) receiving chronic hemodialysis.

The overall objectives are to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of ISIS 416858 in ESRD patients on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease maintained on outpatient hemodialysis at a healthcare center for > 3 months from screening with hemodialysis using heparin (unfractionated heparin or low-molecular weight heparin) 3 times per week for a minimum of 3 hours per dialysis session and plan to continue this throughout the study.

Exclusion Criteria:

* Documented thrombotic event (acute coronary syndrome, stroke or transient ischemic attack, venous thromboembolic event) in the past 3 months.
* Active bleeding within the past 3 months from screening or documented bleeding diathesis (history of bleeding disorder) or Screening values of:

  * Platelet count < 150,000 cells/mm3
  * INR > 1.4
  * aPTT > upper limit of normal (ULN)
* Abnormal liver function at Screening:

  * ALT or AST > 2 x ULN
  * Total bilirubin > ULN
* Concomitant medication restrictions: Concomitant use of anticoagulant/antiplatelet agents (e.g., dabigatran, rivaroxaban, clopidogrel) that may affect coagulation (except low dose aspirin (≤ 100 mg/day) during Treatment and Post-treatment Evaluation Periods is not allowed.
* Uncontrolled hypertension as judged by the Investigator. Patients with a pre- or post-dialysis blood pressure (BP) that is > 160 mmHg on at least 3 of last 5 dialysis treatments.
* Planned major surgery in the next 6 months (e.g. renal transplant surgery)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability - evaluated by reviewing frequency and severity of Adverse events (including bleeding events) and use of concomitant medications, changes in vital signs and laboratory evaluations for all patients | For the PK Cohort: Patients will be followed for 72 days. For Cohorts A and B: Patients will be followed for 162 days.
  The safety and tolerability of ISIS 416858 will be evaluated by reviewing frequency and severity of Adverse events (including bleeding events) and use of concomitant medications, changes in vital signs and laboratory evaluations for all patients

SECONDARY OUTCOMES:
Pharmacodynamic Outcomes in FXI antigen and activity as measured by absolute change over time. | For the PK Cohort: Patients will be followed for 72 days. For Cohorts A and B: Patients will be followed for 162 days.
  Pharmacodynamic Outcomes as measured by absolute change over time for FXI antigen and activity (units/milliliter)
Pharmacodynamic Outcomes in FXI antigen and activity as measured by percent change over time. | For the PK Cohort: Patients will be followed for 72 days. For Cohorts A and B: Patients will be followed for 162 days.
  Pharmacodynamic Outcomes as measured by percent change over time for FXI antigen and activity (units/milliliter)
Pharmacodynamic Outcomes in aPTT as measured by absolute change over time. | For the PK Cohort: Patients will be followed for 72 days. For Cohorts A and B: Patients will be followed for 162 days.
  Pharmacodynamic Outcomes as measured by absolute change over time for aPTT (seconds)
Pharmacodynamic Outcomes in aPTT as measured by percent change over time. | For the PK Cohort: Patients will be followed for 72 days. For Cohorts A and B: Patients will be followed for 162 days.
  Pharmacodynamic Outcomes as measured by percent change over time for aPTT (seconds)
Pharmacodynamic Outcomes for PT and the PT derived INR as measured by absolute change over time. | For the PK Cohort: Patients will be followed for 72 days. For Cohorts A and B: Patients will be followed for 162 days.
  Pharmacodynamic Outcomes as measured by absolute change over time for PT (seconds) and the PT derived INR (International Normalization Ratio)
Pharmacodynamic Outcomes for PT and the PT derived INR as measured by percent change over time. | For the PK Cohort: Patients will be followed for 72 days. For Cohorts A and B: Patients will be followed for 162 days.
  Pharmacodynamic Outcomes as measured by percent change over time for PT (seconds) and the PT derived INR (International Normalization Ratio)

OTHER OUTCOMES:
Pharmacokinetic Outcome for PK Cohort of effect of dialysis on peak concentrations | Patients will be followed for 29 days for this outcome measure.
  Effect of dialysis on peak concentrations post single dose drug administration.
Pharmacokinetic Outcome for PK Cohort of effect of dialysis on partial area under the plasma concentration-time curve | Patients will be followed for 29 days for this outcome measure.
  Effect of dialysis on partial area under the plasma concentration-time curve post single dose drug administration (AUC 0-24hr).
Pharmacokinetic Outcome for Cohorts A and B to assess steady state concentrations | Patients will be followed for 162 days for this outcome measure
  Plasma will be collected at each dosing interval to assess steady state concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Bhanot, MD, Study Director — Ionis Pharmaceuticals
Locations (6):
- Canada (6):
  - Ionis Investigative Site, Edmonton, Alberta
  - Ionis Investigative Site, Halifax, Nova Scotia
  - Ionis Investigative Site, Hamilton, Ontario
  - Ionis Investigative Site, London, Ontario
  - Ionis Investigative Site, Toronto, Ontario
  - Ionis Investigative Site, Montreal, Quebec

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] Walsh M, Bethune C, Smyth A, Tyrwhitt J, Jung SW, Yu RZ, Wang Y, Geary RS, Weitz J, Bhanot S; CS4 Investigators. Phase 2 Study of the Factor XI Antisense Inhibitor IONIS-FXIRx in Patients With ESRD. Kidney Int Rep. 2021 Nov 24;7(2):200-209. doi: 10.1016/j.ekir.2021.11.011. eCollection 2022 Feb. PMID 35155859